CLINICAL TRIAL: NCT03365583
Title: Comparison of Gut Microbial Composition in Breastfed Infants With and Without Vitamin B12 Deficiency
Brief Title: The Impact of Vitamin B12 Deficiency on Infant Gut Microbiota
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2016.137
Record Dates: First submitted 2017-12-02; First posted 2017-12-07 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Vitamin B 12 Deficiency
Keywords: Vitamin B12; Microbiome; infant
MeSH Terms: conditions — Vitamin B 12 Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fecal samples of breastfed infants will be extracted for DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vitamin B12 deficiency: No intervention will be administered for this study. Serum vitamin B12 <203 pg/mL is considered as vitamin B12 deficiency.
  Fecal microbiota composition will be analyzed with 16S rRNA sequencing. In a subgroup of infants (n=11), fecal samples will be recollected after the treatment as usual
- Vitamin B12 sufficient: Serum vitamin B12 ≥203 pg/mL is considered as vitamin B12 sufficient Fecal microbiota composition will be analyzed with 16S rRNA sequencing.

SUMMARY:
Vitamin B12 plays important roles in DNA synthesis and neurological functions. Vitamin B12 deficiency is one of the most common micronutrient deficiencies and it has become increasingly more frequent in infants. The deficiency develops more often between 4 to 12 months of age, coinciding with the decreased fetal storage. The highest rates of vitamin B12 deficiency were observed among infants who are breastfed by mothers receiving a diet low in vitamin B12.

The main objective of this study is to compare the gut microbial composition of healthy term exclusively breastfed infants with or without vitamin B12 deficiency. We hypothesized that gut microbiome differs between vitamin B12 deficient and control infants; pathogenic bacteria are hypothesized to be higher, and beneficial bacteria to be lower in vitamin B12 deficient infants as compared to control.

An observational study in the Marmara University Pendik Research and Training Hospital well child outpatient clinic is conducted in 90 infants. Participants aged between 4 to 6 months who fulfill the inclusion criteria are enrolled.

Inclusion criteria are term birth (>37 gestational weeks), birth weight >2500 gr, absence of congenital anomalies, hemoglobin ≥10 g/dL, and exclusive breastfeeding.

Exclusion criteria include prematurity, low birth weight, intrapartum antibiotic use, current or previous use of infant formula, malnutrition, use of iron supplements, infant use of antibiotics, use of probiotics within the last 8 weeks before study entry, and introduction to solid foods.

Primary outcome measures:Microbial counts, and a comparison of type and abundance of species (predominant, pathogenic, and opportunistic bacteria, yeast, and parasites) between vitamin B12 deficient and sufficient subjects will be assessed.

Secondary outcome measures: Fecal bacterial communities will be assessed before and after treatment in a subgroup of infants.

Each stool sample is collected from cloth diapers, and placed in sterile collection tubes. Samples are kept at 4 C and in less than 5 hours, they are frozen at -80 C until further analysis. Specimens are transported on dry ice to the Diagen Inc for DNA extraction.

For the extraction protocol, QuickGene (Kurabo, North America) extraction device will be used.

The extracted DNA samples will be sent to Diversigen Inc (Houston, USA) for analysis. Fecal microbiota composition will be analyzed with 16S ribosomal ribonucleic acid (rRNA) sequencing.

DETAILED DESCRIPTION:
Vitamin B12 plays important roles in DNA synthesis and neurological functions. Vitamin B12 deficiency is one of the most common micronutrient deficiencies and it has become increasingly more frequent in infants. The deficiency develops more often between 4 to 12 months of age, coinciding with the decreased fetal storage. The highest rates of vitamin B12 deficiency were observed among infants who are breastfed by mothers receiving a diet low in vitamin B12. The data on prevalence of vitamin B12 deficiency in Turkey mainly relate to pregnant women and varies between 34% to 72%. In our previous study, 36.3% of the infants (n=222) were vitamin B12 deficient. The prevalence was even higher (43%) in infants exclusively breastfed for 6 months.

The physiologic and neurologic consequences of micronutrient deficiencies have been addressed extensively. Although it is known that individuals with high bacterial loads in their small intestines tend to have low cobalamin status, less is known about its effects on the developing gut microbiota. It is suggested that early environmental factors influencing gut microbiota during this crucial developmental period can lead to long term consequences on health and disease. The data available is mostly limited to the effects of iron. The review of the literature has not yielded any study, which investigates the effects of vitamin B12 on the developing gut microbiota.

The study is conducted at Marmara University well child outpatient clinic. The clinic is hospital based and located in Pendik, Istanbul. The outpatient clinic provides well child care; and besides anthropometric measurements, infants are routinely screened for anemia at 4 to 6 months of age.

Ninety-two exclusively breastfed infants are approached for eligibility. Two infants are excluded due to prior antibiotic use and 90 infants are enrolled.

Fecal collection tubes are given to the parents of infants who fulfill the inclusion criteria during routine blood withdrawal. For the reporting, serum vitamin B12 <203 pg/mL is considered as vitamin B12 deficiency, and ≥203 pg/mL as vitamin B12 sufficient.

Infants with vitamin B12 deficiency are treated with intramuscular vitamin b12 (hydroxycobalamin), 250-500 mcg twice weekly for a week, and then 500 mcg weekly for another 3 weeks. One month after the supplementation in the recommended dose, stools are recollected in a subgroup of subjects (n=11) with vitamin B12 deficiency.

Samples are kept at 4 C and in less than 5 hours, they are frozen at -80 C until further analysis.

Questionnaires are completed, antropometric measures are taken and fecal samples are transported on dry ice to the Diagen Inc for DNA extraction DNA extraction will be performed by Diagen Inc. For the extraction protocol, QuickGene (Kurabo, North America) extraction device will be used.

The extracted DNA samples will be sent to Diversigen Inc (Houston, USA) for 16S rRNA Gene V4 region sequencing.

ELIGIBILITY:
Inclusion Criteria:

* must be >37 gestational weeks, birth weight must be >2500 gr, must be exclusively breastfed there should be no congenital anomalies, hemoglobin should be ≥10 g/dL,

Exclusion Criteria:

* prematurity, low birth weight, intrapartum antibiotic use, current or previous use of infant formula, malnutrition, use of iron supplements, use of antibiotics, use of probiotics within the last 8 weeks before study entry, and being introduced to solid foods

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy term exclusively breastfed infants aged between 4 to 6 months who fulfill the inclusion criteria are enrolled
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-09-03 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
Gut microbial community differences between infants with vitamin B12 deficiency and infants with sufficient vitamin B12 | DNA extraction and fecal microbiota composition with 16S rRNA sequencing is anticipated to be completed at June 2018
  Microbial counts, and a comparison of type and abundance of species (predominant, pathogenic, and opportunistic bacteria, yeast, and parasites) between vitamin B12 deficient and sufficient subjects will be assessed

SECONDARY OUTCOMES:
Gut microbial community differences within subject | Recollection of stool samples one month after treatment as usual. DNA extraction and fecal microbiota composition with 16S rRNA sequencing is anticipated to be completed at June 2018
  Fecal bacterial communities will be assessed before and after treatment as usual in a subgroup of vitamin B12 deficient infants

CONTACTS AND LOCATIONS:
Overall Officials: Perran Boran, MD, PhD, Principal Investigator — Marmara University
Locations (1):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)